CLINICAL TRIAL: NCT06740838
Title: Overnight Dexamethasone in Primary Aldosteronism Screening in Patients on Interfering Therapy (the ODEPRASC Study)
Brief Title: Overnight Dexamethasone in Primary Aldosteronism Screening
Acronym: ODEPRASC
Status: Recruiting | Type: Observational
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Sponsor
Other Study IDs: NKBBN 287-76/2021
Record Dates: First submitted 2024-12-14; First posted 2024-12-18 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2024-12

CONDITIONS: Primary Aldosteronism; Hypertension
Keywords: primary aldosteronism; screening; renin; aldosterone; hypertension; corticotropin; dexamethasone
MeSH Terms: conditions — Hyperaldosteronism; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Post-DXM ARR development cohort: Data from the first half of participants data will be used to generate post-DXM ARR (and possibly Ald) thresholds, which will be subsequently temporally validated in the confirmatory cohort.
- Post-DXM ARR confirmatory cohort: Post-DXM ARR thresholds will be applied among participants of the confirmatory cohort, however, these will also undergo the medication withdrawal, OSLT, and other PA confirmatory tests if indicated.

SUMMARY:
The goal of this observational study is to learn whether screening for primary aldosteronism can be improved among patients on chronic blood pressure-lowering medications by ordering intake of 1 mg of dexamethasone prior to hormonal examinations.

Primary aldosteronism is a condition, in which an adrenal gland steroid aldosterone is released in excessive amounts; it commonly causes hypertension but requires specific therapy different from usually prescribed in other forms of hypertension.

Dexamethasone is a synthetic steroid used for both therapeutic and diagnostic purposes. A single 1 mg dexamethasone dose taken at 11 p.m. in order to measure hormone concentrations the following morning (so called overnight 1-mg dexamethasone test) is a commonly applied test in the work-up of adrenal disorders.

The main question the project aims to answer is:

Can screening for primary aldosteronism be improved among patients receiving blood pressure-lowering medications with overnight 1-mg dexamethasone intake?

Participants will undergo changes in their chronic medication to be able to definitely rule out or confirm primary aldosteronism in blood hormonal examinations. These modifications and modifications are not part of the research project.

For this project participants will be asked to

* undergo the 1-mg dexamethasone test one to three times in order to compare hormonal concentrations before and after it,
* collect urine for 24 hours to determine aldosterone in the urine sample after medications interfering in aldosterone release are temporarily withdrawn.

DETAILED DESCRIPTION:
Background Primary aldosteronism (PA) underlies or contributes to hypertension (HT) in up to 30% of patients. In the last two decades PA has been demonstrated to encompass mild forms, which do not meet established diagnostic criteria, yet are still clinically relevant. However, PA has been shown to be vastly underdiagnosed: less than 5% of patients from at-risk populations undergo screening.

One of the main reasons for low PA screening prevalence is the recommendation of hypotensive therapy modification prior to hormonal assessment, i.e. withdrawal of medications interfering in the renin-angiotensin-aldosterone system (RAAS) (2016 Endocrine Society guideline, 2020 European Society of Hypertension consensus statement). On the other hand, in many instances, PA may be diagnosed despite treatment with RAAS-interfering drugs.

Previous research showed efficacy in the diagnostic approach toward PA can be greatly improved by incorporating adrenocorticotropic hormone (ACTH) suppression. This was achieved by determining PA screening and confirmatory thresholds following a 2-day 2-mg/day dexamethasone (DXM) test. Patients diagnosed with PA by meeting these novel diagnostic criteria responded well to mineralocorticoid receptor antagonists.

These two diagnostic approaches (work-up in patients receiving RAAS-interfering drugs along with ACTH suppression) have not been combined so far.

Aim To generate and temporally validate PA screening thresholds (aldosterone-to-renin ratio, ARR, and aldosterone, Ald) among patients with HT receiving medications interfering in the RAAS by applying overnight ACTH suppression.

Methodology The project received the consent of the local bioethics committee. A development cohort of n=80, and a confirmation cohort of n=80, amount to 240 participants total due to an expected withdrawal rate of 33%. Study participants will be enrolled in a single, tertiary-care endocrine hospital in one-day clinic setting among hypertensive patients undergoing hormonal examinations due to the presence of an adrenocortical lesion with radiological features of an adenoma or hyperplasia (ACA or AHA, respectively). Only patients with indications for further PA testing upon a positive, permissive ARR will be recruited for participation in the study. Further diagnostic procedures (both in the course of this research and clinically-indicated) will be conducted in an outpatient endocrine clinic. Exclusion criteria include non-viability for RAAS-interfering medication modification.

Basal (1) ARR will be required for inclusion, while in the course of the project participants will undergo ARR measurements post-DXM on own (chronic) medications (2), pre- and post-DXM ARR upon partial modification of RAAS-interfering medications (3 and 4), and pre- and post-DXM upon temporary withdrawal of RAAS-interfering medications (5 and 6). An oral salt loading test, OSLT (one of established confirmatory PA tests), will be performed off interfering medications in all patients. Also, patients with a positive PA screening result will undergo either seated saline-infusion (SIT) and/or captopril challenge test (CCT) to confirm PA in a one-day clinic. Results of these confirmatory tests will be used as reference in determining sensitivity and specificity of PA screening thresholds on RAAS-interfering therapy regimens.

Statistical analysis will be performed upon gathering clinical and hormonal data to determine thresholds for ARR, aldosterone and renin to suggest optimal (simple but more accurate than currently applied) PA screening criteria.

Expected results The hypotheses of the project are

1. Eliminating the effect of ACTH on Ald release will result in better interpretability of ARR and/or renin and Ald thresholds, and
2. Complete withdrawal of RAAS-interfering medications is not required for PA screening upon ARR determination combined with ACTH suppression.

The objective of the study is demonstrating that ARR measurement following overnight 1-mg DXM intake reduces the equivocal rate in interpreting the ARR measurement in PA screening compared to conventional ARR.

ELIGIBILITY:
Inclusion Criteria:

* suspected or diagnosed HT,
* age between 40 and 75,
* available aldosterone and renin result at the time of one-day clinic stay,
* scheduled 1-mg-DXM test (indicated for possible mild autonomous cortisol secretion, MACS),
* presence of an adrenal lesion with radiologic features of adrenocortical adenoma/hyperplasia.

Exclusion Criteria:

* baseline (pre-DXM) hyperreninemia (renin exceeding the upper limit of normal at the study site, i.e. 46.1 mIU/l, assay manufacturer: Diasorin),
* baseline (pre-DXM) Ald<3 ng/dl,
* overt clinical and/or biochemical features of adrenal hormone deficiency or excess other than MACS (8 a.m. cortisolemia in the 50-140 nmol/l range in the 1-mg DXM test),
* therapy with glucocorticoids, non-steroidal anti-inflammatory drugs, hormonal replacement therapy, hormonal contraceptive therapy, and/or licorice intake,
* established or suspected secondary HT other than due to PA,
* comorbidities including: poorly controlled and/or other than type 2 diabetes mellitus (T2DM), present and past alcohol abuse, obesity grade 3 (i.e. body mass index of at least 40 kg/m2), severe CV disease disqualifying a patient from chronic medication modification, active malignancy, decompensated autoimmune disease as well as an autoimmune disease associated with cardiovascular and/or renal complications, estimated glomerular filtration rate (eGFR) below 45 ml/min/1.73m2, poor physical condition, lack and withdrawal of consent for participation.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * patients of the one-day endocrine clinic of the Department of Endocrinology and Internal Medicine of the University Clinical Center of the Medical University of Gdansk, admitted for hormonal work-up due to an adrenal lesion,
  * study design is cross-sectional
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Overall diagnostic accuracy of post-DXM ARR | 24 months
  percentage of correctly categorized patients with hypertension on RAAS-interfering medications as either with clear or unclear PA screening threshold base on post-DXM ARR determination

SECONDARY OUTCOMES:
Association between post-DXM ARR and 24-h urinary aldosteronuria in the oral salt loading test | 24 months
  Post-DXM ARRs on different medications will be investigated for correlations or other associations with urinary aldosteronuria in the OSLT.

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Kmiec, MD, Ph.D., Principal Investigator — Department of Endocrinology and Internal Medicine, Medical University of Gdansk
Locations (1):
- Department of Endocrinology and Internal Medicine, University Clinical Center, Medical University of Gdansk, Gdansk, Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No
IRB approval and participant consent do not cover sharing IPD outside the scope of the study.

REFERENCES:
- [Background] Upton TJ, Zavala E, Methlie P, Kampe O, Tsagarakis S, Oksnes M, Bensing S, Vassiliadi DA, Grytaas MA, Botusan IR, Ueland G, Berinder K, Simunkova K, Balomenaki M, Margaritopoulos D, Henne N, Crossley R, Russell G, Husebye ES, Lightman SL. High-resolution daily profiles of tissue adrenal steroids by portable automated collection. Sci Transl Med. 2023 Jun 21;15(701):eadg8464. doi: 10.1126/scitranslmed.adg8464. Epub 2023 Jun 21. PMID 37343084
- [Background] Yozamp N, Hundemer GL, Moussa M, Underhill J, Fudim T, Sacks B, Vaidya A. Intraindividual Variability of Aldosterone Concentrations in Primary Aldosteronism: Implications for Case Detection. Hypertension. 2021 Mar 3;77(3):891-899. doi: 10.1161/HYPERTENSIONAHA.120.16429. Epub 2020 Dec 7. PMID 33280409
- [Background] Markou A, Sertedaki A, Kaltsas G, Androulakis II, Marakaki C, Pappa T, Gouli A, Papanastasiou L, Fountoulakis S, Zacharoulis A, Karavidas A, Ragkou D, Charmandari E, Chrousos GP, Piaditis GP. Stress-induced Aldosterone Hyper-Secretion in a Substantial Subset of Patients With Essential Hypertension. J Clin Endocrinol Metab. 2015 Aug;100(8):2857-64. doi: 10.1210/jc.2015-1268. Epub 2015 May 14. PMID 25974737
- [Background] Papanastasiou L, Markou A, Pappa T, Gouli A, Tsounas P, Fountoulakis S, Kounadi T, Tsiama V, Dasou A, Gryparis A, Samara C, Zografos G, Kaltsas G, Chrousos G, Piaditis G. Primary aldosteronism in hypertensive patients: clinical implications and target therapy. Eur J Clin Invest. 2014 Aug;44(8):697-706. doi: 10.1111/eci.12286. PMID 24909545
- [Background] Gouli A, Kaltsas G, Tzonou A, Markou A, Androulakis II, Ragkou D, Vamvakidis K, Zografos G, Kontogeorgos G, Chrousos GP, Piaditis G. High prevalence of autonomous aldosterone secretion among patients with essential hypertension. Eur J Clin Invest. 2011 Nov;41(11):1227-36. doi: 10.1111/j.1365-2362.2011.02531.x. Epub 2011 May 3. PMID 21534948
- [Background] Markou A, Kaltsas GA, Papanastasiou L, Gravvanis C, Voulgaris N, Kanti G, Zografos GN, Chrousos GP, Piaditis G. Enhanced performance of a modified diagnostic test of primary aldosteronism in patients with adrenal adenomas. Eur J Endocrinol. 2022 Jan 6;186(2):265-273. doi: 10.1530/EJE-21-0625. PMID 34882580
- [Background] Li X, Liang J, Hu J, Ma L, Yang J, Zhang A, Jing Y, Song Y, Yang Y, Feng Z, Du Z, Wang Y, Luo T, He W, Shu X, Yang S, Li Q; Chongqing Primary Aldosteronism Study (CONPASS) Group. Screening for primary aldosteronism on and off interfering medications. Endocrine. 2024 Jan;83(1):178-187. doi: 10.1007/s12020-023-03520-6. Epub 2023 Oct 5. PMID 37796417
- [Background] Seifarth C, Trenkel S, Schobel H, Hahn EG, Hensen J. Influence of antihypertensive medication on aldosterone and renin concentration in the differential diagnosis of essential hypertension and primary aldosteronism. Clin Endocrinol (Oxf). 2002 Oct;57(4):457-65. doi: 10.1046/j.1365-2265.2002.01613.x. PMID 12354127
- [Background] Browne GA, Griffin TP, O'Shea PM, Dennedy MC. beta-Blocker withdrawal is preferable for accurate interpretation of the aldosterone-renin ratio in chronically treated hypertension. Clin Endocrinol (Oxf). 2016 Mar;84(3):325-31. doi: 10.1111/cen.12882. Epub 2015 Sep 22. PMID 26300226
- [Background] Brown JM, Robinson-Cohen C, Luque-Fernandez MA, Allison MA, Baudrand R, Ix JH, Kestenbaum B, de Boer IH, Vaidya A. The Spectrum of Subclinical Primary Aldosteronism and Incident Hypertension: A Cohort Study. Ann Intern Med. 2017 Nov 7;167(9):630-641. doi: 10.7326/M17-0882. Epub 2017 Oct 10. PMID 29052707
- [Background] Parksook WW, Brown JM, Omata K, Tezuka Y, Ono Y, Satoh F, Tsai LC, Niebuhr Y, Milks J, Moore A, Honzel B, Liu H, Auchus RJ, Sunthornyothin S, Turcu AF, Vaidya A. The Spectrum of Dysregulated Aldosterone Production: An International Human Physiology Study. J Clin Endocrinol Metab. 2024 Aug 13;109(9):2220-2232. doi: 10.1210/clinem/dgae145. PMID 38450549
- [Background] McEvoy JW, McCarthy CP, Bruno RM, Brouwers S, Canavan MD, Ceconi C, Christodorescu RM, Daskalopoulou SS, Ferro CJ, Gerdts E, Hanssen H, Harris J, Lauder L, McManus RJ, Molloy GJ, Rahimi K, Regitz-Zagrosek V, Rossi GP, Sandset EC, Scheenaerts B, Staessen JA, Uchmanowicz I, Volterrani M, Touyz RM; ESC Scientific Document Group. 2024 ESC Guidelines for the management of elevated blood pressure and hypertension. Eur Heart J. 2024 Oct 7;45(38):3912-4018. doi: 10.1093/eurheartj/ehae178. No abstract available. PMID 39210715
- [Background] Mulatero P, Sechi LA, Williams TA, Lenders JWM, Reincke M, Satoh F, Januszewicz A, Naruse M, Doumas M, Veglio F, Wu VC, Widimsky J. Subtype diagnosis, treatment, complications and outcomes of primary aldosteronism and future direction of research: a position statement and consensus of the Working Group on Endocrine Hypertension of the European Society of Hypertension. J Hypertens. 2020 Oct;38(10):1929-1936. doi: 10.1097/HJH.0000000000002520. PMID 32890265
- [Background] Mulatero P, Monticone S, Deinum J, Amar L, Prejbisz A, Zennaro MC, Beuschlein F, Rossi GP, Nishikawa T, Morganti A, Seccia TM, Lin YH, Fallo F, Widimsky J. Genetics, prevalence, screening and confirmation of primary aldosteronism: a position statement and consensus of the Working Group on Endocrine Hypertension of The European Society of Hypertension. J Hypertens. 2020 Oct;38(10):1919-1928. doi: 10.1097/HJH.0000000000002510. PMID 32890264
- [Background] Funder JW, Carey RM, Mantero F, Murad MH, Reincke M, Shibata H, Stowasser M, Young WF Jr. The Management of Primary Aldosteronism: Case Detection, Diagnosis, and Treatment: An Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2016 May;101(5):1889-916. doi: 10.1210/jc.2015-4061. Epub 2016 Mar 2. PMID 26934393
- [Background] Vaidya A, Carey RM. Evolution of the Primary Aldosteronism Syndrome: Updating the Approach. J Clin Endocrinol Metab. 2020 Dec 1;105(12):3771-83. doi: 10.1210/clinem/dgaa606. PMID 32865201
- [Background] Brown JM, Siddiqui M, Calhoun DA, Carey RM, Hopkins PN, Williams GH, Vaidya A. The Unrecognized Prevalence of Primary Aldosteronism: A Cross-sectional Study. Ann Intern Med. 2020 Jul 7;173(1):10-20. doi: 10.7326/M20-0065. Epub 2020 May 26. PMID 32449886
- [Background] Funder JW. Who and How Should We Screen for Primary Aldosteronism? Hypertension. 2023 Dec;80(12):2495-2500. doi: 10.1161/HYPERTENSIONAHA.123.20536. Epub 2023 Oct 6. PMID 37800386
- [Derived] Kmiec P, Okroj D, Zdrojewska M, Fiszer J, Zembrzuska S, Swiatkowska-Stodulska R. Overnight Dexamethasone in Primary Aldosteronism Screening in Patients on Interfering Therapy (ODEPRASC): A Diagnostic Interpretability Study Protocol. J Clin Hypertens (Greenwich). 2025 Nov;27(11):e70180. doi: 10.1111/jch.70180. PMID 41268804